CLINICAL TRIAL: NCT02710890
Title: A Multicenter, Open-Label Study to Investigate the Safety and Tolerability of Intravenous Lacosamide in Children (>= 1 Month to < 17 Years of Age) With Epilepsy
Brief Title: Study to Investigate Safety and Tolerability of Intravenous Lacosamide in Children.
Acronym: ASPIRE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0060; 2014-003294-42 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2016-03-09; First posted 2016-03-17 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2020-11

CONDITIONS: Epilepsy
Keywords: Epilepsy; pediatric; intravenous; children; Lacosamide; VIMPAT®; seizure
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lacosamide (Experimental): Up to 2 age-based Cohorts with Cohort 1 including at least 40 subjects who are >=8 to <17 years. For Cohort 2 every attempt will be made to enroll 20 subjects >= 4 to < 8 years of age, 12 subjects >= 2 to < 4 years of age and 12 subjects >= 1 month to < 2 years of age. A Data Monitoring Committee (DMC) will review the safety and tolerability data for each Cohort to make the following recommendations: the progression of the current Cohort, including intravenous (iv) infusion durations to be evaluated, and progression to initiate enrollment in the next Cohort (Cohort 2).
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Pharmaceutical form: solution for infusion
  Concentration: 10 mg/ml
  Route of Administration: intravenous
  Other Names: Vimpat

SUMMARY:
EP0060 is a multicenter, open-label study to evaluate the safety and tolerability of intravenous (iv) Lacosamide (LCM) in pediatric subjects >= 1 month to < 17 years of age with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from >=1 month to <17 years of age
* Subject has a diagnosis of epilepsy with partial-onset seizures or primary generalized tonic-clonic seizures
* Subject meets 1 of the following criteria:

  1. Open-label lacosmide (OLL) subject: Subject is currently receiving oral lacosmide (LCM) as adjunctive or monotherapy as participants in an open label long-term study (SP848, EP0034, or other pediatric study); OR,
  2. Prescription lacosamide (RxL) subject: Subject is currently receiving prescribed oral LCM from commercial supply (eg, VIMPAT) as adjunctive or monotherapy; OR,
  3. Initiating intravenous lacosamide (IIL) subject: Subject is not currently receiving LCM and will receive intravenous (iv) LCM as adjunctive treatment in EP0060. Initiation of LCM monotherapy is not permitted in IIL subjects.
* Subject is an OLL or RxL subject and meets both of the following criteria:

  1. Subject has been administered LCM for the treatment of epilepsy for at least 2 weeks prior to Screening; AND
  2. Subject has been administered (OLL) or prescribed (RxL) oral LCM at a dose of 2 mg/kg/day to 12 mg/kg/day (for subjects <50 kg) or 100 mg/day to 600 mg/day (for subjects >=50 kg). Open-label study drug LCM (OLL) or prescribed oral LCM dose (RxL) must be stable for at least 3 days prior to first LCM infusion; OR,
* Subject is an ILL subject and is on a stable dosage regimen of at least 1 antiepileptic drug (AED). The daily dosage regimen of concomitant AED therapy must be kept constant for a period of at least 2 weeks prior to Screening.
* Subject is an acceptable candidate for venipuncture and iv infusion
* Subject is, in the opinion of the investigator, able to comply with all study requirements. Subject (or parent[s] or legal representative) is willing to comply with all study requirements
* Subject weighs >=4 kg

Exclusion Criteria:

* Subject has previously received intravenous (iv) lacosamide (LCM) in this study
* Subject has any medical, neurological, or psychiatric condition that, in the opinion of the investigator, could jeopardize the subject's health or compromise the subject's ability to participate in EP0060
* Subject has clinically significant hypotension or bradycardia in the opinion of the investigator
* Subject >=6 years of age has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by positive responses ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening

For open-label lacosamide (OLL) subjects, enrollment in EP0060 is not permitted if any of the following additional criteria are met:

- Subject has any ongoing Adverse Event (AE) in their long-term, open-label study that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate EP0060 or the subject meets any of the criteria for required withdrawal from the long-term open-label study

For prescription lacosamide (RxL) and initiating intravenous lacosamide (IIL) subjects, enrollment in EP0060 is not permitted if any of the following additional criteria are met:

* Subject has a medical condition that could reasonably be expected to interfere with drug absorption distribution, metabolism, or excretion
* Subject is a female of childbearing potential and does not practice an acceptable method of contraception for the duration of participation in EP0060
* Subject has creatinine clearance less than 30 mL/min
* Subject has a clinically relevant electrocardiogram (ECG) abnormality, in the opinion of the principal investigator (ie, second or third degree heart block at rest or a QT prolongation greater than 450 ms)
* Subject has hemodynamically significant heart disease (eg, heart failure)
* Subject has an arrhythmic heart condition requiring medical therapy, known cardiac sodium channelopathy, such as Brugada syndrome
* Subject has a known history of severe anaphylactic reaction or serious blood dyscrasias
* Subject has an acute or subacutely progressive central nervous system disease.
* Subject has epilepsy secondary to a progressing cerebral disease or any other progressive or neurodegenerative disease (malignant brain tumor or Rasmussen syndrome)
* Lacosamide is intended for treatment of generalized convulsive status epilepticus
* Subject has diagnosis of Dravet's syndrome

For IIL subjects, enrollment in EP0060 is not permitted if the following additional criterion is met:

- Subject has been treated with LCM within the last 3 months prior to Screening

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 8445992273 (UCB)
Locations (23):
- United States (10):
  - Ep0060 003, Birmingham, Alabama
  - Ep0060 010, Little Rock, Arkansas
  - Ep0060 008, Loxahatchee Groves, Florida
  - Ep0060 009, Saint Paul, Minnesota
  - Ep0060 014, Henderson, Nevada
  - Ep0060 002, New Brunswick, New Jersey
  - Ep0060 006, Akron, Ohio
  - Ep0060 011, Cincinnati, Ohio
  - Ep0060 005, Dallas, Texas
  - Ep0060 007, San Antonio, Texas
- Hungary (2):
  - Ep0060 400, Budapest
  - Ep0060 401, Debrecen
- Italy (3):
  - Ep0060 503, Messina
  - Ep0060 505, Roma
  - Ep0060 502, Verona
- Ep0060 701, Krakow, Poland
- Ukraine (7):
  - Ep0060 224, Dnipro
  - Ep0060 225, Dnipro
  - Ep0060 220, Ivano-Frankivsk
  - Ep0060 221, Kiev
  - Ep0060 222, Kiev
  - Ep0060 226, Kiev
  - Ep0060 223, Vinnytsia

REFERENCES:
- [Result] Farkas MK, Beller C, Bozorg A, McClung C, Roebling R, Yates T, Yuen N, Makedonska I. Safety and tolerability of short-term infusions of intravenous lacosamide in pediatric patients with epilepsy: An open-label, phase 2/3 trial. Epilepsia Open. 2023 Mar;8(1):146-153. doi: 10.1002/epi4.12682. Epub 2023 Jan 18. PMID 36529709
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in May 2017 and concluded in June 2019.
Pre-assignment Details: Participant Flow refers to the Safety Set iv (SS-iv).
Groups:
- Lacosamide Age Cohort ≥ 1 Month - < 8 Years: This arm consisted of participants who formed Cohort 2, were greater than or equal to (≥) 1 month to less than (<) 8 years of age and received at least 1 dose of intravenous (iv) lacosamide (LCM). For the first 20 participants in Cohort 2, iv LCM has been infused over a duration of 30 minutes but no longer than 60 minutes whenever possible. After completion of the first 20 participants in Cohort 2, a Data Monitoring Committee (DMC) reviewed the safety and tolerability data for this Cohort and made the following recommendations: the progression of the current Cohort, including iv infusion durations to be evaluated.
- Lacosamide Age Cohort ≥ 8 - < 17 Years: This arm consisted of participants who formed Cohort 1, were ≥ 8 to < 17 years of age and received at least 1 dose of iv LCM. For the first 20 participants in Cohort 1, iv LCM has been infused over a duration of 30 minutes but no longer than 60 minutes whenever possible. After completion of the first 20 participants in Cohort 1, a DMC reviewed the safety and tolerability data for this Cohort and made the following recommendations: the progression of the current Cohort, including iv infusion durations to be evaluated, and progression to initiate enrollment in the next Cohort (Cohort 2).
Period: Overall Study
Arm/Group | Lacosamide Age Cohort ≥ 1 Month - < 8 Years | Lacosamide Age Cohort ≥ 8 - < 17 Years
Started | 48 | 55
Completed | 48 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Safety Set iv (SS-iv) which consisted of study participants in the Safety Set (SS) who received at least 1 dose of EP0060 study medication intravenous (iv) lacosamide (LCM)
Arm/Group | Lacosamide Age Cohort ≥ 1 Month - < 8 Years | Lacosamide Age Cohort ≥ 8 - < 17 Years | Total Title
Number analyzed (Participants) | 48 | 55 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 55 | 103
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.840 (2.329) | 12.662 (2.409) | 8.551 (5.013)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 31 | 57
  Male | 22 | 24 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black | 2 | 3 | 5
  White | 46 | 50 | 96
  Other/Mixed | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Adverse Event Reported Spontaneously by the Participant/or Caregiver (Including Parent/Legal Guardian) or Observed by the Investigator During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  26 adverse events are reported splitting into at least 19 occurrences of individual pre-treatment emergent adverse events and 7 treatment emergent adverse events (TEAEs).
Time Frame: From Screening Period (Day -7 to Day -1) up to the End-of-Study Period (up to Day 37)
Population: The Safety Set iv (SS-iv) included study participants in the Safety Set (SS) who received at least 1 dose of EP0060 study medication iv LCM.
Measure: Number; unit: percentage of participants
Groups:
- Lacosamide Age Cohort ≥ 1 Month - < 8 Years (SS-iv): This arm consisted of participants who formed Cohort 2, were ≥ 1 month to < 8 years of age and received at least 1 dose of iv LCM. For the first 20 participants in Cohort 2, iv LCM has been infused over a duration of 30 minutes but no longer than 60 minutes whenever possible. After completion of the first 20 participants in Cohort 2, a DMC reviewed the safety and tolerability data for this Cohort and made the following recommendations: the progression of the current Cohort, including iv infusion durations to be evaluated. Participants formed the Safety Set iv (SS-iv).
- Lacosamide Age Cohort ≥ 8 - < 17 Years (SS-iv): This arm consisted of participants who formed Cohort 1, were ≥ 8 to < 17 years of age and received at least 1 dose of iv LCM. For the first 20 participants in Cohort 1, iv LCM has been infused over a duration of 30 minutes but no longer than 60 minutes whenever possible. After completion of the first 20 participants in Cohort 1, a DMC reviewed the safety and tolerability data for this Cohort and made the following recommendations: the progression of the current Cohort, including iv infusion durations to be evaluated, and progression to initiate enrollment in the next Cohort (Cohort 2). Participants formed the Safety Set iv (SS-iv).
Arm/Group | Lacosamide Age Cohort ≥ 1 Month - < 8 Years (SS-iv) | Lacosamide Age Cohort ≥ 8 - < 17 Years (SS-iv)
Number analyzed (Participants) | 48 | 55
percentage of participants | 12.5 | 14.5

2. Primary Outcome: Percentage of Participants That Withdrew Due to Adverse Events During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment and led to the withdrawal of the participants from the study. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Screening Period (Day -7 to Day -1) up to the End-of-Study Period (up to Day 37)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide Age Cohort ≥ 1 Month - < 8 Years (SS-iv) | Lacosamide Age Cohort ≥ 8 - < 17 Years (SS-iv)
Number analyzed (Participants) | 48 | 55
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were reported from Visit 2/Day 1 until End of Study Period (29 to 37 days after Visit 2/Day 1).
Description: 1 participant could experience multiple adverse events.
Arm/Group | Lacosamide Age Cohort ≥ 1 Month - < 8 Years (SS-iv) | Lacosamide Age Cohort ≥ 8 - < 17 Years (SS-iv)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/55
Other Adverse Events (participants affected / at risk) | 3/48 | 2/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide Age Cohort ≥ 1 Month - < 8 Years (SS-iv) (N=48) | Lacosamide Age Cohort ≥ 8 - < 17 Years (SS-iv) (N=55)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT02710890/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT02710890/SAP_000.pdf